CLINICAL TRIAL: NCT06364423
Title: Phase I/II Trial of Anti-CD19 Chimeric Antigen Receptor T-Cell Immunotherapy for Chronic Lymphocytic Leukemia (CLL)
Brief Title: Anti-CD19 Chimeric Antigen Receptor T-Cell Immunotherapy for Chronic Lymphocytic Leukemia (CLL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001599; 001599-C
Record Dates: First submitted 2024-04-12; First posted 2024-04-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; B-Lymphocytic Leukemia, Chronic
Keywords: Chimeric Antigen Receptors; Autologous T Cells Infusion; Adoptive T Cell Therapy; Gene Therapy; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; Immunotherapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Rituximab, conditioning chemotherapy plus CAR T-cells- Dose escalation (Experimental): Escalating dose of anti-CD19 CAR T- cells/kg + rituximab and conditioning chemotherapy
  Interventions: Biological: Autologous HuCD19 ( Anti-CD19)CAR T cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab
- 2/Rituximab, conditioning chemotherapy plus CAR T-cells- Dose expansion (Experimental): MTD dose or Optimal dose of Anti-CD19 CAR T- cells/kg + rituximab and conditioning chemotherapy
  Interventions: Biological: Autologous HuCD19 ( Anti-CD19)CAR T cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Biological: Autologous HuCD19 ( Anti-CD19)CAR T cells — 1.0x10^6 CAR+T-cells - 12x10^6 CAR+ T cells/kg (weight based dosing per cohort) infused on day 0
Drug: Cyclophosphamide — 500 mg/m^2 IV infusion over 30 minutes on days -5, -4 and -3
Drug: Fludarabine — 30 mg/m^2 IV infusion over 30 minutes administered immediately following the cyclophosphamide on days -5, -4,and -3
Drug: Rituximab — 500 mg/m2 IV infusion over 30 minutes on day -5; 375 mg/m2 IV infusion over 30 minutes on days 2-9 prior to apheresis

SUMMARY:
Background:

Chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) are blood cancers that affect certain white blood cells. Advanced forms of these diseases are difficult to treat. CD19 is a protein often found on the surfaces of these cancer cells. Researchers can modify a person's own immune cells (T cells) to target CD19. When these modified T cells are returned to the body-a treatment called anti-CD19 chimeric antigen receptor (CAR) T cell therapy-they may help kill cancer cells.

Objective:

To test anti-CD19 CAR T cell therapy in people with CLL or SLL.

Eligibility:

People aged 18 years and older with CLL or SLL that has not been controlled with standard drugs.

Design:

Participants will be screened. They will have imaging scans and tests of their heart function. If a sample of tissue from their tumor is not available, a new one may be taken; the sample will be tested for CD19.

Participants will receive a drug to reduce the leukemia cells in their blood. Then they will undergo apheresis: Blood will be taken from the body through a needle. The blood will pass through a machine that separates out the T cells. The remaining blood will be returned to the body through a different needle. The collected T cells will be gene edited to make them attack cells with CD19.

Participants will take drugs to prepare them for treatment for 3 days. These drugs will start 5 days before the treatment. Then their own modified CAR T cells will be returned to their bloodstream. Participants will stay in the hospital for at least 9 days after the treatment.

Follow-up visits will continue for 5 years.

DETAILED DESCRIPTION:
Background:

* Improved treatments for relapsed and refractory chronic lymphocytic leukemia (CLL) are needed.
* T cells can be genetically modified to express chimeric antigen receptors (CARs) that specifically target malignancy-associated antigens.
* Autologous T cells genetically modified to express CARs targeting the B-cell antigen CD19 have caused complete remissions in patients with leukemia or lymphoma. However, there is no FDA-approved CAR T-cell product for CLL. Responses to CAR T-cell therapy in CLL have historically been lower than in other B-cell malignancies.
* CD19 is uniformly expressed on CLL.
* CD19 is not expressed by normal cells except for B cells, follicular dendritic cells, and some plasma cells.
* We have constructed a novel gene therapy construct that encodes a fully-human anti-CD19 CAR.
* The conditioning regimen for this trial will include rituximab, fludarabine, and cyclophosphamide.
* Possible toxicities include cytokine-associated toxicities such as fever, hypotension, and neurological toxicities. Elimination of normal B cells is probable, and unknown toxicities are also possible.

Primary objective, Phase I:

-Determine the safety of administering a novel conditioning regimen and T cells expressing the Hu19-CD828Z CAR to participants with advanced CLL.

Primary objective, Phase II:

-Determine the overall response rate (ORR) of a novel conditioning regimen and T cells expressing the Hu19-CD828Z CAR for participants with advanced CLL.

Eligibility:

* Participant must have CLL or small lymphocytic lymphoma (SLL).
* Age >= 18 years of age
* Participant must have malignancy that is measurable on a CT scan or by flow cytometry of bone marrow or blood.
* Participant must have a creatinine of 1.5 mg/dL or less and a normal cardiac ejection fraction.
* An ECOG performance status of 0-1 is required.
* No active infections are allowed including hepatitis B or hepatitis C.
* Absolute neutrophil count >= 1000/microL, platelet count >= 50,000/microL, hemoglobin >= 8g/dL
* Serum ALT and AST less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated.
* At least 14 days must elapse between the time of any prior systemic treatment (including corticosteroids) and the first dose of protocol-required rituximab. In addition, 60 days must elapse from therapy with antibody-based treatments targeting CD19 and CAR T-cell infusion.
* Prior CAR T-cell therapy is not allowed.
* Demonstration of CD19 expression by the CLL/SLL is required for eligibility.
* CD19 expression must be uniform . Uniform CD19 expression is defined as no obvious CD19-negative CLL/SLL being present.

Design:

* This is a phase I dose-escalation trial with an expansion cohort (Phase II portion)
* T cells obtained by leukapheresis will be genetically modified to express the Hu19-CD828Z CAR.
* Participants will receive 2 doses of rituximab and a lymphocyte-depleting chemotherapy conditioning regimen with the intent of decreasing the burden of CLL, which might reduce toxicity and improve anti-leukemia outcomes.
* Rituximab will be given in 2 doses, of 375 mg/m^2 for the first dose and 500 mg/m^2 for the second dose.
* The chemotherapy conditioning regimen is cyclophosphamide 500 mg/m^2 daily for 3 days and fludarabine 30 mg/m^2 daily for 3 days. Fludarabine will be given on the same days as the cyclophosphamide.
* Three days after the chemotherapy ends, participants will receive an infusion of CAR T cells.
* The initial dose level of this dose-escalation trial will be 1.0x10^6 CAR+ T cells/kg of recipient bodyweight.
* The CAR T-cell cell dose administered will be escalated until a maximum tolerated dose or an optimal dose is determined.
* Following the T-cell infusion, there is a mandatory 9-day inpatient hospitalization to monitor for toxicity.
* Outpatient follow-up is planned for 2 weeks and 1, 2, 3, 4, 6, 9, and 12 months after the CAR T-cell infusion; less frequent follow-up is required more than 1 year after infusion. Long-term gene-therapy follow-up for a total of 15 years after infusion is required.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Malignancy criteria

  * Histologically confirmed participants with either CLL or SLL will be eligible.
  * Demonstration of CD19 expression on CLL/SLL, as assessed by the NCI Laboratory of Pathology or NIH Department of Laboratory Medicine Hematopathology section.
  * CD19 expression must be uniform meaning no populations of clearly CD19-negative CLL/SLL cells are observed.
  * Participants must have received prior systemic therapy. The last dosage of systemic therapy (including corticosteroids) must be at least 14 days prior to the first dose of rituximab.
  * For participants who have received antibodies targeting CD19, at least sixty days must elapse between therapy with antibodies targeting CD19 and CAR T-cell infusion.
  * Participants must have received at least two prior treatment regimens at least one of which must have contained a Bruton s tyrosine kinase (BTK) inhibitor. Participants who took a BTK inhibitor but stopped due to intolerance are potentially eligible.
  * All participants must have measurable malignancy as defined by at least one of the criteria below.

    * Presence of CLL or SLL masses that are measurable (minimum 1.5 cm in largest diameter) by CT scan is required unless bone marrow or blood involvement with malignancy is detected. All masses must be less than or equal to 10.0 cm in the largest diameter.
    * For CLL with only bone marrow and/or blood involvement, no mass is necessary, but if a mass is not present, bone marrow and/or blood malignancy must be detectable by flow cytometry. Any level of CLL detectable by flow cytometry is sufficient.
* Other inclusion criteria:

  * Age >= 18 years.
  * Performance status (ECOG) 0-1.
  * Participants must have adequate organ and marrow function as defined below:

    * ANC >= 1,000/mcL without the support of filgrastim or other growth factors in the 10 days prior to screening assessment
    * platelets >= 50,000/mcL without transfusion support
    * hemoglobin >= 8 g/dL
    * total bilirubin <= 2.0 mg/dL
    * ALT or AST Serum ALT and AST less or equal to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated. If liver involvement with malignancy is detected, ALT and AST must be less than or equal to 5 times the upper limit of normal
    * Serum Creatinine Serum creatinine levels < 1.5 X institutional ULN. Participants with serum creatinine >= 1.5 X institutional ULN may participate if serum creatinine eGFR is >=50 mL/min/1.73m^2 by 2021 CKD-EPI equation.

      * ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);
      * AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.
      * (A)Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard.
  * B cells must make up less than 90% of blood lymphocytes on a lymphocyte phenotyping profile TBNK at the time of screening assessment.
  * Room air oxygen saturation of 92% or greater
  * Participants of child-bearing or child-fathering potential must be willing to practice abstinence or highly effective contraception starting at the time of study entry, for the duration of study therapy, and for 12 months after receiving the protocol treatment, or until CAR T cells are no longer detectable in the blood, whichever is later.
  * Participants must agree not to donate eggs for 12 months after receiving the protocol treatment, or until CAR T cells are no longer detectable in the blood, whichever is later.
  * Participants who are breastfeeding must be willing to cease breastfeeding from study treatment initiation through 6 months after the last dose of the study drug(s), or until CAR T cells are no longer detectable in the blood, whichever is later.
  * Participants must have a negative blood PCR test for hepatitis B DNA. If hepatitis B DNA (PCR) testing is not available, participants must have a negative hepatitis B surface antigen and negative hepatitis B core antibody test.
  * Participants must have a negative blood PCR test for hepatitis C RNA. Only if Hepatitis C PCR testing is not available in a timely manner, participants must have a negative Hepatitis C antibody test.
  * Cardiac ejection fraction of greater than or equal to 50% by echocardiography and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 30 days prior to treatment start.
  * All participants must have the ability to understand and willingness to sign a written informed consent.
  * All participants must be willing to undergo mandatory biopsies during the study. A bone marrow biopsy will be required prior to the chemotherapy and CAR T-cell infusion. Another bone marrow biopsy will be required approximately 14 days after CAR T-cell infusion.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents.
* Participants who have had prior CAR T-cell therapy.
* Participants who have had a live-attenuated or viral vector-based vaccine in the last 60 days prior to pre-leukapheresis rituximab. Participants who plan to receive a live attenuated or viral vector-based vaccine within the first 100 days after CAR T-cell infusion.
* Participants that require urgent therapy due to tumor mass effects or spinal cord compression.
* Participants that have active hemolytic anemia.
* Current/active HIV infection, as measured by seropositivity for HIV antibody.
* Participants with second malignancies in addition to their CLL are not eligible if the second malignancy has required treatment with surgery, radiation or chemotherapy, or other therapies within the past 3 years or is not in complete remission. Exceptions are that, in the last 3 years, participants may have had successful resection of nonmetastatic basal cell or squamous cell carcinoma of the skin, and participants may have received hormonal therapy for fully resected breast cancer.
* Positive beta Human chorionic gonadotropin (Beta-HCG) serum or urine pregnancy test in women of childbearing potential (WOCBP) performed at screening.
* Active uncontrolled systemic infections (defined as infections causing fevers within 48 hours of the date of planned protocol rituximab or chemotherapy start and infections requiring intravenous antibiotics when intravenous antibiotics have been administered for less than 72 hours at the time of protocol rituximab or chemotherapy start). There must be objective evidence of infection, including, but not limited to, a positive blood, urine or sputum culture, positive nasal swab or blood test for viral infection, or the appearance of infiltrates on imaging of the lung.
* Active coagulation disorders or other major uncontrolled medical illnesses of the cardiovascular, respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system, history of myocardial infarction, history of ventricular tachycardia or ventricular fibrillation, active cardiac arrhythmias (Resolved atrial fibrillation that is not treated with anticoagulants is allowed.), active obstructive or restrictive pulmonary disease, active autoimmune diseases such as rheumatoid arthritis.These include uncontrolled intercurrent illness manifesting as electrolyte derangements or as assessed by chemistries.
* Significant neurologic disorders, including a history of a seizure disorder as an adult, that are not completely and permanently resolved and not requiring current treatment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Prior allogeneic stem cell transplant
* Systemic corticosteroid steroid therapy of any dose greater than 5 mg/day or more of prednisone or equivalent is not allowed within 14 days prior to the first dose of rituximab. Corticosteroid creams, ointments, and eye drops are allowed.
* Participants on systemic anticoagulant therapy except aspirin.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study, including hypersensitivity to aminoglycoside antibiotics, which may be used in the cell culture media.
* Active central nervous system/brain metastases or cerebrospinal fluid malignancy.
* Checkpoint inhibitor drugs such as pembrolizumab or nivolumab or other antibodies targeting PD-1 or PDL-1 within 180 days of pre-leukapheresis rituximab. This is because of possible effects checkpoint inhibitor therapy could have on the participant's T cells.
* Known active alcohol or drug abuse.
* History of allergy to study drug components.
* Active tumor lysis syndrome as assessed by serum uric acid, LDH, calcium, and phosphorus.
* Active rhabdomyolysis as assessed by elevated CK and acute change in renal function as reflected by increased creatinine and blood urea nitrogen (BUN).
* Active diabetic ketoacidosis or hyperosmolar hyperglycemic state, as assessed by serum glucose. The urine will be tested for ketones if serum glucose is over 350 mg/dL at screening.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determine the safety of administering T-cells expressing a fully-human anti-CD19 CAR to participants with advanced CLL or SLL. | From time of the pre-leukapheresis rituximab through 5 years after CAR T infusion.
  Adverse Events (AE) by type, grade, and frequency
Phase II: Determine the overall response rate (ORR) of T cells expressing an anti-CD19 CAR with a fully-human single chain variable fragment (scFv) to participants with advanced CLL | From time of the pre-leukapheresis rituximab through 5 years after CAR T infusion.
  Overall Response Rate will be evaluated using published criteria; these will be reported along with a 95% confidence interval

SECONDARY OUTCOMES:
Phase I: Assess overall response rate | up to 5 years
  Overall Response rate (ORR= CR + PR) will be recorded if ORR occurs at any response assessment time-point.
Phase I+II: Assess complete response rate | up to 5 years
  Complete Response rate (CR) in participants who receive subsequent infusion, up to 5 years after entry date for last participant
Phase I+II: Assess duration of responses | up to 5 years
  Duration of response from date of response will be measured for no more than 5 years after the last participant has been enrolled on the trial.
Phase I+II: Determine the ORR for re treatment with rituximab, chemotherapy and CAR T cells in eligible patients | up to 5 years
  Overall Response rate (ORR= CR + PR) for re-treatment with Rituximab will be recorded if ORR occurs at any response assessment time-point.
Phase II: Determine the frequency of grade 3-4 adverse events at the Optimal Dose | up to 5 years
  Adverse Events (AE) by type, grade, and frequency

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.@@@@@@This study will comply with the NIH Genomic Data Sharing (GDS) Policy, which applies to all new and ongoing NIH IRP-funded research, as of January 25, 2015, that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001599-C.html